CLINICAL TRIAL: NCT03481764
Title: Anthropogenetic Variability in the Group of Individuals With Febrile Seizures - Population Genetic Study
Brief Title: Anthropogenetic Variability in the Group of Individuals With Febrile Seizures
Status: Completed | Type: Observational
Sponsor: Institut za Rehabilitaciju Sokobanjska Beograd (Other)
Responsible Party: Principal Investigator, Tamara Filipovic, Principal Investigator, Institut za Rehabilitaciju Sokobanjska Beograd
Other Study IDs: Sbcprn
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Febrile Seizure
Keywords: febrile seizure; HRC-test; genetic variation; epilepsy
MeSH Terms: conditions — Seizures, Febrile; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- FS: Febrile Seizures: Involved patient with diagnosed Febrile Seizures which were hospitalized or recieved ambulatory treatment in University Children´s Hospital in Belgrade. Ages 5-14 years
  Interventions: Genetic: HRC-test
- CN: Control group: The control group was made of healthy children older than 5 years of age, which have never had any neurological disorders in their anamnesis and who were patients in preschool or school dispensaries in the city of Belgrade
  Interventions: Genetic: HRC-test
- SFS : group of individuals with simple FS: Simplex febrile seizures (SFS) last shorter than 15 minutes and their type is tonic-clonic. Also, they did not show signs of recidivism during the first 24 hours and were diagnosed at the patients aged from 6th months to 5th year
  Interventions: Genetic: HRC-test
- CFS : group of individuals with complex FS: Complex febrile seizures (CFS) were diagnosed at those patients that had focal seizure or epileptic status or seizure having the body temperature lower than 38 degree, which occurred outside of the typical age group and finally which repeated in the first 24 hours again
  Interventions: Genetic: HRC-test
- WFS: group of individuals with FS and without epilepsia: group of children with Febrile Seizure and not developed epilepsia
  Interventions: Genetic: HRC-test
- EFS: group of individuals with epilepsia and Febrile Seizures: Group of children with Febrile Seizures, who have developed Epilepsy
  Interventions: Genetic: HRC-test

INTERVENTIONS:
Genetic: HRC-test — Using HRC-test we analyze 20 selected genetically controlled morphophysiological traits among FS children and control.Homozygous-recessive traits in the region of human head are: attached ear lobe,continuous frontal hair line,blue eyes straight hair,soft hair and blond hair,double hair whorl,hair whorl orientation-opposite from clock-wise,as well as an inability to roll,fold and curve the tongue,a guttural "r and Daltonism.HRC trait expressed in human arms and legs, such as distal or proximal hyper-extensibility of the thumb,index finger shorter than the ring finger,left-handedness, hand clasping pattern.In order to achieve high level of objectivity during the process of data gathering, the same person conducting all testing.Inside the group of charcteristics which show high level of variability,only the extreme phenotypes were considered recessive.For the purpose of testing the color blindness in examinees,the Pseudoisochromatic plates test was used.

SUMMARY:
Febrile seizures(FS) are the most common neurological disorder in chilhood and are a great stress for parents due to their dramatic clinical appearance.

Using HRC-test(test for determination of homozygously recessive characteristics in humans) we analyzed presence, distribution, and individual combination of 20 selected genetically controlled morpho-physiological traits among FS patients and control to determine a possible deviation in the homozygosity level and genetic loads in the group of affected children and whether there is a predisposition to the occurrence of FS.

DETAILED DESCRIPTION:
Febrile seizures(FS) are one of the most common neurological disorders in children and infants. It is estimated that 2-5% of children younger than 5 years of age experience at least one epileptic seizure during the period of febrile seizure.

FS, as defined by the American Academy of Pediatrics (AAP), are " seizure occurring in febrile children between the ages of 6 and 60 months who do not have an intracranial infection, metabolic disturbance, or history of afebrile seizures ".

The diagnosis of FS is based on physical examination and anamnesis taken from the gardian, aiming primarily to detect the real cause that led to a FS.

The etiology of FS is complex and it is still the subject of numerous studies and research done in the field. However, there is strong evidence showing that heterogeneous genetic predisposition interacting with various risk factors can lead to a FS.

There are several risk factors mentioned in literature which can cause the first FS. One of the most important is positive family history of FS (especially among the closest relatives) . Other possible factors include: high body temperature (the higher level of body temperature increases the risk of a seizure occurrence), preexisting neurodevelopment delay , neonatal care longer that 28 days.

The development of epilepsy after FS moves around 3%, after simple febrile seizure (SFS) the risk is around 2% whereas after complex febrile seizure (CFS) it is about 2 to 3%. Around 13% of epilepsy patients have experienced FS once. Prolonged FS can lead to mesial temporal sclerosis and to temporal lobe epilepsy, but the level of risk is still uncertain.

The research shows that abnormal neurological development before the FS, the occurrences of a febrile seizures among relatives, as well as the CFS, represent risk factors for emergence of epilepsy after the FS.

Since FS are genetically controlled, it is presumed that increased homozygosity and decreased variability in patients can be in correlation with the expression of FS.

The determination of the presence of homozygous-recessive characteristics (HRC) in individuals with FS provides an insight whether the prevalence of homozygous or heterozygous loci on different chromosomes exists. The number of homozygous recessive traits represent one type of indicator of the homologous chromosomal homozygosity, which can vary significantly both at the individual, as well as at the group level.

ELIGIBILITY:
Inclusion Criteria:

* Our research has involved patient with diagnosed Febrile Seizure which were hospitalized or recieved ambulatory treatment in University Children´s Hospital in Belgrade.

Exclusion Criteria:

* Patients with evidence of intracranial infections
* Patients with incomplited medical documentation

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The Febrile Seizure affected children as well as the individuals from the control group were members of the same population (Serbian)
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
To establish the degree of genetic homozygosity and variability in subjects with Febrile Seizure and control group | 2 years
  Using HRC-test (test for determination of homozygously recessive characteristics in humans) we will analyzed presence, distribution, and individual combination of 20 selected genetically controlled morpho-physiological traits among FS patients and control to determine a possible deviation in the homozygosity level and genetic loads in the group of affected children and whether there is a predisposition to the occurrence of FS.

SECONDARY OUTCOMES:
Establish a correlation between the degree of genetic homozygosity and variability between subjects with SFS and CFS, also WFS and EFS | 2 years
  The results of HRC test shows a degree of genetic homozygosity as well as the level of possible genetic loads what may indicate to the presence of genetic problems which further affect the capacity of normal development, with the possibility for more extreme cases to develop specific properties including increased or desreased resistance to certain types of illness

CONTACTS AND LOCATIONS:
Locations (1):
- Sanja Dimitrijevic, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Nikolic D, Petronic I, Cvjeticanin S, Brdar R, Cirovic D, Bizic M, Konstantinovic L, Matanovic D. Gender and morphogenetic variability of patients with spina bifida occulta and spina bifida aperta: prospective population-genetic study. Hippokratia. 2012 Jan;16(1):35-9. PMID 23930055
- [Background] Cvjeticanin S, Marinkovic D. Morphogenetic variability during selection of elite water polo players. J Sports Sci. 2009 Jul;27(9):941-7. doi: 10.1080/02640410902960494. PMID 19629843
- [Background] Marinkovic D, Cvjeticanin S. Population-genetic study of Balkan endemic nephropathy in Serbia. Genetika. 2007 Aug;43(8):1134-8. PMID 17958315
- [Background] Cvjeticanin S, Marinkovic D. Genetic variability in the group of patients with congenital hip dislocation. Genetika. 2005 Aug;41(8):1142-6. PMID 16161637
- [Background] Khair AM, Elmagrabi D. Febrile Seizures and Febrile Seizure Syndromes: An Updated Overview of Old and Current Knowledge. Neurol Res Int. 2015;2015:849341. doi: 10.1155/2015/849341. Epub 2015 Nov 30. PMID 26697219
- [Background] Dimitrijevic S, Cvjeticanin S, Pusica A, Jekic B, Filipovic T, Nikolic D. Anthropogenetic Variability in the Group of Individuals with Febrile Seizures: Population-Genetic Study. Biomed Res Int. 2018 Jul 5;2018:7845904. doi: 10.1155/2018/7845904. eCollection 2018. PMID 30069480